CLINICAL TRIAL: NCT05136274
Title: Evaluation of Ipsilateral Tubal Patency After Conservative Medical or Surgical Treatment in Uncomplicated Ectopic Pregnancy, "Hospital General", Angola 2021-2022
Brief Title: Evaluation of Ipsilateral Tubal Patency After Conservative Medical or Surgical Treatment.
Acronym: EENCBE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: EDGREM Investimentos (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Eduardo Kedisobua, Medical Surgery, EDGREM Investimentos
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDINV-EENC
Record Dates: First submitted 2021-11-08; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Ectopic Pregnancy
Keywords: uncomplicated ectopic pregnancy methotrexate
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial comparing ipsilateral tubal patency with the use of two therapeutic methods, groups A; with intramuscular methotrexate administration and B conservative surgery (linear salpingostomy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical treatment (Active Comparator): By administering a single intramuscular dose of 50mg / m2 / Sc of Methotrexate.
  Interventions: Drug: Medical treatment
- Surgical treatment (Active Comparator): Will be performed by laparoscopy or laparotomy, using the Linear Salpingostomy technique.
  Interventions: Drug: Medical treatment

INTERVENTIONS:
Drug: Medical treatment — The surgical treatment group can be laparoscopically or by laparotomy, using the Linear Salpingostomy technique. Follow-up with β fraction of chorionic gonadotropin on days 0, 3, 7 and 14 together with gynecological abdominal or transvaginal ultrasound on day 0 and 7 and hysterosalpingography will be performed after three months of treatment.
  Other Names: Surgical treatment

SUMMARY:
Ectopic Pregnancy is an entity in which a fertilized ovum is implanted outside its normal place, is considered a public health problem worldwide and is one of the main causes of maternal mortality in the first trimester. The availability of high sensitivity methods of detection of gonadotrophins and the use of high resolution transvaginal ultrasonography have allowed an earlier diagnosis of the same, enabling less aggressive treatments such as the use of parenteral MTX, with the intention of avoiding mutilating surgical treatment , preserving the tube and eventually improving future fertility expectations. The surgical treatment is of choice, this can be laparoscopically or by laparotomy. In this case, we need to preserve fertility, the most indicated is linear salpingostomy; In spite of the existence other techniques.

DETAILED DESCRIPTION:
The EP constitutes a frequent obstetric emergency in Angola and the province of Benguela is not exempt from this health problem. Every day we see women with this pathology, to which, most of them, they undergo a mutilating surgical treatment (salpingectomy) that impedes their future reproductive capacity. The procreation in the African continent and especially in Angola, has great social and family implications that can reach the breaking of marriages and family (broadcast and study of the Public Television of Angola in the program "Na lente" no year 2018 Taking into account the importance of procreation in the welfare and stability of the marital relationship.Main Objectiv: To demonstrate the non-inferiority of conservative treatment with MTX in ipsilateral tubal patency after an uncomplicated ectopic pregnancy compared with surgical treatment with linear salpingostomy in the Hospital General, Angola

ELIGIBILITY:
Inclusion Criteria:

Patient presenting with Ectopic Pregnancy, associated with quantitative titers of βHCG ≥ 100 mUI / ml, without intrauterine gestational sac.

Patient presenting uncomplicated Ectopic Pregnancy with an adnexal mass diameter ≤4 cm diagnosed by abdominal and / or transvaginal ultrasonography.

Absence of heartbeat. No toxicity to MTX. Normal laboratory tests (blood count, coagulogram, liver and kidney function). Hemodynamic stability.

Exclusion Criteria:

* Complicated Ectopic Pregnancy.
* Ectopic pregnancy is out of the tuba on ultrasound
* Patients with Immunosuppression.
* Allergy to MTX.
* Patients with Active Respiratory Disease, Blood Dyspasia, Peptic Ulcer, Renal Insufficiency and Hepatic Insufficiency.
* Do not accept to participate in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 204 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-08-17 (Estimated); Study Completion 2023-08-17 (Estimated)

PRIMARY OUTCOMES:
Incidence of Ipsilateral tubal patency | A hysterosalpingography will be performed 3 months after the treatment.
  Incidence of Ipsilateral tubal patency

SECONDARY OUTCOMES:
Incidence of Achieve the gestation and the culmination. | Up to two years
  Incidence of Achieve the gestation and the culmination.

CONTACTS AND LOCATIONS:
Overall Officials: Moreno Araujo, Study Chair — EDGREN INVESTIMENTOS
Locations (1):
- Maria Dolores Reguera Saborido, Benguela, Angola